CLINICAL TRIAL: NCT03770104
Title: Correct Endotracheal Tube Position in Newborns Intubated in the Delivery Room According to Two Different Methods Based on Estimated Birth Weight. Randomized Clinical Trial (NeoTEDI)
Brief Title: Correct Endotracheal Tube Position in Newborns Intubated in the Delivery Room
Acronym: Intubated-DR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tania Carbayo Jiménez (Other)
Responsible Party: Sponsor-Investigator, Tania Carbayo Jiménez, Tania Carbayo Jimenez, MD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Neo TEDI
Record Dates: First submitted 2018-12-05; First posted 2018-12-10 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Intubation Complication; Newborn Morbidity; Cardiopulmonary Resuscitation
Keywords: Intubation; Newborn; Delivery room; Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinicians and neonatal nurses will not masked to group assignment. However, Neonatal Intensive Care Unit nurses who take care of the patient will be mask, as well as both pediatric radiologist who will determine the main outcome of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (5.5 plus weight) (Experimental): ETT insertion depth using Spanish recommendations Patients included in the intervention group arm who are included in the study will be intubated using Spanish recommendations (5.5 plus weight) to estimate insertion endotracheal tube depth. In addition, every arm will be divided into 2 subgroups depending on gestational age (under 32 weeks or equal/over 32 weeks' gestation).
  Interventions: Procedure: ETT insertion depth using Spanish recommendations
- Control Group (6 plus weight) (Experimental): ETT insertion depth using international recommendations Patients included in the intervention group arm who are included in the study will be intubated using international recommendations (6 plus weight) to estimate insertion endotracheal tube depth. In addition, every arm will be divided into 2 subgroups depending on gestational age (under 32 weeks or equal/over 32 weeks' gestation).
  Interventions: Procedure: ETT insertion depth using international recommendations

INTERVENTIONS:
Procedure: ETT insertion depth using Spanish recommendations — Infants included in this assignment group will be intubated using the formula 5.5 plus weight, when requiring oral intubation in the delivery room.
  Arms: Intervention Group (5.5 plus weight)
Procedure: ETT insertion depth using international recommendations — Infants included in this assignment group will be intubated using the formula 6 plus weight, when requiring oral intubation in the delivery room.
  Arms: Control Group (6 plus weight)

SUMMARY:
The investigators wished to determine whether estimating endotracheal tube (ETT) insertion depth using the formula given by Spanish guidelines recommendations (5,5 plus weight) rather than the depth using the formula given by international guidelines recommendations (6 plus weight) resulted in more correctly positioned endotracheal tube tips in newborns intubated in the delivery room.

DETAILED DESCRIPTION:
A number of different methods have been used to guide clinicians in estimating the correct depth of insertion of endotracheal tube (ETT) at the time of oral intubation. Minor differences in tube length may lead to intubation of the right main bronchus or extubation. However, none of them has shown to be better than others when compared in the context of randomized clinical trials.

Commonly, clinicians use a formula based on the newborn's weight (Tochen formula: ETT insertion depth (cm)=6 + wt (kg)). While this method is widely used and recommended by international guidelines, it has been found to frequently result in incorrectly positioned tubes, especially in infants <1000 g in weight in whom it may lead to overestimation of ETT insertion depth.

On the other hand, Spanish Society of Neonatology recommended in their last published guidelines (2017) to use an alternative version formula (ETT insertion depth (cm)=5.5 + wt (kg)), which is commonly used among Spanish neonatal units.

Finally, no studies have been performed in newborns who require oral intubation in the delivery room, since these intubations are usually excluded because infants are not routinely weighed prior to resuscitation and weight can not be rapidly obtained. Given that Obstetric Unit in our hospital is a high standard one with a highly reliable estimated fetal weight in prenatal ultrasound, the investigators will use estimated fetal weight referred on ultrasounds or 50th percentile for gestational age for calculations.

ELIGIBILITY:
Inclusion Criteria:

* All newborns requiring endotracheal oral intubation in the delivery room after birth.
* Parents accept deferred informed consent to participate in the study.

Exclusion Criteria:

* Prior to randomization
* Uncontrolled gestation where both estimated fetal weight and gestational age are unknown.
* Upper airway anomaly or a lung anomaly that would distort the upper airway anatomy.
* Infants who require nasotracheal intubation
* Infants who are intubated in the Neonatal Intensive Care Unit
* Post-randomization
* Newborns who are randomized but finally do not require intubation
* Intubated newborns who are electively extubated in the delivery room
* Parents / legal guardian refuse to give consent to participate in the study

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of correct endotracheal tube (ETT) position | 1 hour
  Correct ETT position, that is, tip between the upper border of the first thoracic vertebra (T1) and the lower border of the second thoracic vertebra (T2) on a chest X-ray as determined by one pediatric radiologist masked to group assignment.

SECONDARY OUTCOMES:
Number of intubation attempts in the delivery room | 2 days
  Number of intubation attempts in the delivery room by healthcare professionals
Number of accidental extubations prior to chest X-ray | 2 days
  Number of accidental extubations prior to chest X-ray confirmation of ETT position
Frequency of ETT repositioning prior and after chest X-ray | 2 days
  ETT repositioning prior and after chest X-ray
Frequency of incorrect ETT position | 2 days
  Incorrect ETT position (too low or too high)
Frequency of complications secondary to incorrect ETT position | 7 days
  Complications secondary to incorrect ETT position (air leak, unplanned extubation, atelectasis)
Professional healthcare sensation about correct or incorrect ETT position | 1 day
  Professional healthcare sensation about correct or incorrect ETT position, before confirmation with Chest X-ray confirmation
Duration of ventilation | 3 months
  Duration of ventilation in days
Oxygen therapy at 28 days | 1 month
  Oxygen therapy at 28 days
Oxygen therapy at 36 weeks postmenstrual age | 3 months
  Oxygen therapy at 36 weeks postmenstrual age

OTHER OUTCOMES:
Presence of intraventricular hemorrhage or central nervous system lesion | 3 months
  Presence of intraventricular hemorrhage or central nervous system lesion
Death before discharge from the hospital | 4 months
  Death before discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Tania Carbayo Jimenez, M.D., Study Chair — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre. Neonatology Department., Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flinn AM, Travers CP, Laffan EE, O'Donnell CP. Estimating the endotracheal tube insertion depth in newborns using weight or gestation: a randomised trial. Neonatology. 2015;107(3):167-72. doi: 10.1159/000369375. PMID 25592171
- [Background] Gill I, Stafford A, Murphy MC, Geoghegan AR, Crealey M, Laffan E, O'Donnell CPF. Randomised trial of estimating oral endotracheal tube insertion depth in newborns using weight or vocal cord guide. Arch Dis Child Fetal Neonatal Ed. 2018 Jul;103(4):F312-F316. doi: 10.1136/archdischild-2017-312798. Epub 2017 Sep 7. PMID 28883098
- [Background] Tochen ML. Orotracheal intubation in the newborn infant: a method for determining depth of tube insertion. J Pediatr. 1979 Dec;95(6):1050-1. doi: 10.1016/s0022-3476(79)80309-1. No abstract available. PMID 501484
- [Background] Amarilyo G, Mimouni FB, Oren A, Tsyrkin S, Mandel D. Orotracheal tube insertion in extremely low birth weight infants. J Pediatr. 2009 May;154(5):764-5. doi: 10.1016/j.jpeds.2008.11.057. PMID 19364561
- [Background] Peterson J, Johnson N, Deakins K, Wilson-Costello D, Jelovsek JE, Chatburn R. Accuracy of the 7-8-9 Rule for endotracheal tube placement in the neonate. J Perinatol. 2006 Jun;26(6):333-6. doi: 10.1038/sj.jp.7211503. PMID 16642028
- [Background] Kempley ST, Moreiras JW, Petrone FL. Endotracheal tube length for neonatal intubation. Resuscitation. 2008 Jun;77(3):369-73. doi: 10.1016/j.resuscitation.2008.02.002. Epub 2008 Mar 26. PMID 18372092